CLINICAL TRIAL: NCT06554275
Title: CCHS SHARE: A Multi-center Longitudinal Natural History Study
Brief Title: CCHS Secure Health-hub Advancing Research Efforts (CCHS SHARE)
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (AP-HP) : Hôpital de la Pitié-Salpêtrière (Unknown); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Hopital Universitaire Robert-Debre (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-7201; 1R01FD008217-01 (FDA)
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Congenital Central Hypoventilation Syndrome
Keywords: Natural History; Rare Disease
MeSH Terms: conditions — Congenital central hypoventilation syndrome; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to capture longitudinal natural history data in Congenital Central Hypoventilation Syndrome (CCHS). This will include capturing standardized clinical data from standard of care assessments at several CCHS referral centers. Funding source-FDA OOPD

DETAILED DESCRIPTION:
The natural history of a disease is how a disease progresses over time and impacts the lives of patients and their families. In Congenital Central Hypoventilation Syndrome (CCHS), as in all rare diseases, collecting enough information to understand disease natural history is challenging. Knowledge and data sharing is a key to overcoming this challenge. Investigators at Lurie Children's are collaborating with teams at other CCHS medical and research centers and patient advocacy groups to build a shared resource called the CCHS Secure Health-hub Advancing Research Efforts (CCHS SHARE). CCHS SHARE will advance knowledge of CCHS natural history and guide future research studies and clinical trials. The purpose of this study is to collect and store CCHS natural history data over the course of many years in CCHS SHARE. Collected information will include patient and family self-reports surrounding their health and its impact on daily life, information collected during standard clinical care (medical records), family history, and other related information from patients. Information in CCHS SHARE will be used for medical research to better understand CCHS and to develop new treatments.

ELIGIBILITY:
Inclusion Criteria:

Participants with a confirmed CCHS diagnosis (confirmed alveolar hypoventilation and PHOX2B mutation testing results), of all ages and genders, who are followed clinically.

Exclusion Criteria:

An unconfirmed diagnosis of CCHS or unconfirmed PHOX2B mutation or not followed clinically

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any individual with a confirmed CCHS diagnosis treated clinically at any of the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Quality of Life | Up to every 14 months
  Patient reported outcome common data elements reflecting core aspects of CCHS will be captured using the Pediatric Quality of Life Inventory (PedsQL) and the 36-item Short Form Health Survey (SF-36)
Caregiver Burden | Up to every 14 months
  Caregiver burden will be assessed using the Zarit Burden Interview
Patient and Caregiver Sleep | Up to every 14 months
  Patient and caregiver sleep will be assessed using PROMIS Sleep Disturbance and Sleep-Related Impairment short forms
Autonomic Symptom Profile | Up to every 14 months
  Validated measures of autonomic function will be captured including data elements from COMPASS-31 and a patient-reported clinical and disease-specific outcomes symptomatology questionnaire relating to CCHS.
Characterize CCHS from a clinical perspective using standardized common data elements (CDEs) in the clinical setting. | Up to every 14 months
  CDEs will include key data points from standard of care assessments of respiratory and cardiovascular function, sleep, exercise capacity, neurocognition, and blood labs.

CONTACTS AND LOCATIONS:
Overall Officials: Debra E Weese-Mayer, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Maxime Patout, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP) : Hôpital de la Pitié-Salpêtrière; Martin Samuels, MD, Principal Investigator — Great Ormond Street Hospital-London (GOSH); Christophe Delclaux, MD, Principal Investigator — Hopital Universitaire Robert-Debre
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States